CLINICAL TRIAL: NCT00608465
Title: Defining Strategies for Improving Endothelial and Fibrinolytic Dysfunction in Obesity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, James Muldowney, Assistant Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 060369; 060369
Record Dates: First submitted 2008-01-22; First posted 2008-02-06 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Metabolic Syndrome X
Keywords: Fibrolytic Dysfunction; Obesity; PAI-1
MeSH Terms: conditions — Metabolic Syndrome; Obesity | interventions — Eplerenone; Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment A (Active Comparator): Eplerenone (study drug)
  Interventions: Drug: Eplerenone
- Treatment B (Active Comparator): Ramipril
  Interventions: Drug: Ramipril

INTERVENTIONS:
Drug: Eplerenone — 5 mg x 1 week followed by 10 mg x 9 weeks.
  Other Names: Inspra
  Arms: Treatment A
Drug: Ramipril — Ramipril 5mg qd x 1 week f/b Ramipril qd x 9 weeks.
  Arms: Treatment B

SUMMARY:
The combination of high blood pressure and having central obesity is an increasing important factor for heart disease in men and women. It can also lead to the early development of hardening of the arteries and increased risk of a stroke. This study will analyze patients' genetic make up to identify who may be at greater risk for heart disease and strokes in relationship to high blood pressure and central obesity.

DETAILED DESCRIPTION:
Obesity is an increasingly important risk factor for cardiovascular disease in men and women and is associated with the premature development of atherosclerosis, and increased risk of stroke. A classical perspective of cardiovascular risk does not adequately explain all of the cardiovascular events associated with obesity. Elevated plasma levels of plasminogen activator inhibitor type I (PAI-1) are one of the biochemical hallmarks for obesity and likely contribute the increased risk of atherothrombotic events in patients with obesity. The central hypothesis of this proposal is that the increased risk of atherothrombotic events in patients with obesity. The central hypothesis of this proposal is that vascular PAI-1 excess promotes the development of intravascular thrombosis. We will test the hypothesis that secreted factors from adipocytes have autocrine, paracrine and endocrine effects that have a deleterious effect on the fibrinolytic system, either by enhancing PAI-1 production or impairing endothelial t-PA release. From a public health perspective, there is no greater threat to America's cardiovascular health than the epidemic of obesity. It is anticipated that this study will provide new insights nto the molecular mechanisms that contribute to the development of fibrinolytic dysfunction and cardiovascular disease in obesity.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between the ages of 18 to 65 years of age.
* Documented diagnosis for the metabolic syndrome:
* Subjects with hypertension (SP>130mmHg)
* Subjects with central obesity (females waist >35"; males waist >40")
* Subjects with dyslipidemia (HDL <40mg/dl, triglycerides > 150 mg/dl)
* Subjects who are insulin resistance (fasting glucose >100mg/dl)

Exclusion Criteria:

* Subjects who smoke
* Women who are pregnant (confirmed by urine beta-HCG).
* Women who are breast feeding
* Subjects with documentation of the following health risk:

  * Subjects with serum creatinine >2.0 mg/dl (males), >1.8 mg/dl (females)
  * Subjects whose creatinine clearance < 50 mls/min
  * Subjects with serum potassium >5.5mEql
  * Subjects with Type 2 diabetes with microalbuminuria (spot urine protein/creatinine ration >0.2)
* Subjects who are currently taking the following medications:
* Warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-05 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James AS Muldowney, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: The study was never unblinded as enrollment was never completed.
Period: Overall Study
Arm/Group | All Patients
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Secreted Factors From Adipocytes Have Autocrine, Paracrine and Endocrine Effects That Have a Deleterious Effect on the Fibrinolytic System, Either by Enhancing PAI-1 Production or Impairing Endothelial t-PA Release
Time Frame: 10-Week period
Population: Enrollment was never completed so study was never unblinded and data was never analyzed
Arm/Group | All Patients
Number analyzed (Participants) | 0

2. Primary Outcome: This Study Will Analyze Patients' Genetic Make up to Identify Who May be at Greater Risk for Heart Disease and Strokes in Relationship to High Blood Pressure and Central Obesity.
Time Frame: 10-weeks
Population: Enrollment was never completed so study was never unblinded and data was never analyzed
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No